CLINICAL TRIAL: NCT05991700
Title: Anthocyanin-Rich Table Grape Powder for Prophylaxis of Post-Operative Atrial Fibrillation
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: California Table Grape Commission (Other)
Responsible Party: Principal Investigator, Steven Bolling, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00211419
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Post-operative Atrial Fibrillation (POAF)

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Concentrated grape powder (Experimental)
  Interventions: Drug: Freeze-Dried California Table Grape
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Freeze-Dried California Table Grape — Consume 2 servings (30.66g/serving) per day for three days before cardiac surgery
  Arms: Concentrated grape powder
Drug: Placebo — Consume 2 servings (30.66g/serving) per day for three days before cardiac surgery
  Arms: Placebo

SUMMARY:
Postoperative atrial fibrillation (POAF) is a common complication following cardiac surgery and leads to worse outcomes. POAF is thought to be caused by the inflammatory state following cardiac surgery. It may be that anti-inflammatory medications could lower the occurrence of POAF, however many typical anti-inflammatory medications, such as ibuprofen, are contraindicated in the post cardiac surgery patient due to increased risks of bleeding. If a drug was identified with anti-inflammatory properties with minimal deleterious side effects, this could be broadly applied to cardiac surgery patients for the prevention of POAF. Interestingly, several small trials have shown that medications that alter transcription of inflammatory markers lead to decreased POAF. Furthermore, we have shown that phytochemicals, such as those found in grapes, have excellent bioavailability and can affect cardiac gene transcription related to inflammation. In this study, we propose to evaluate the efficacy of preoperative administration of concentrated grape powder in the prevention of POAF.

DETAILED DESCRIPTION:
Voluntary recruitment hold pending approval of new protocol.

ELIGIBILITY:
Inclusion Criteria:

* Males and female patients (age 50-79) at the Mitral Valve Clinic/CVC undergoing elective cardiac surgery for mitral valve repair without the Cox MAZE procedure (MVR patients also undergoing CABG and/or tricuspid valve repair are also eligible)
* In sinus rhythm (no pre-operative atrial fibrillation)

Exclusion Criteria:

* Age ≥ 80 years
* Diagnosed pre-operative chronic or paroxysmal AF
* Prior ablation procedure for AF
* Previous cardiac surgery
* Implanted pacemaker
* Active smoker
* Comorbidities such as congenital or cardiac re-operation
* Use of antiarrhythmic agents
* Active inflammatory or infectious disease or malignancy
* Diagnosed autoimmune disease
* Corticosteroid or other immunomodulatory or immunosuppressive medication
* Risk factors for POAF including low ejection fraction (EF) (EF<50%), left atrial (LA) dilation (LA>5.0 cm), and high degree of mitral regurgitation (grade 3-4).

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
POAF-related events during initial hospital stay and within 30 days after surgery | 30 days
Atrial transcripts related to NFκB activation; Impact on NIDDM, Angiotensin II | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan - Michigan Medicine, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No